CLINICAL TRIAL: NCT01077648
Title: Occurrence of Brain Metastasis in Breast Cancer Patients Diagnosed at Advanced Stages of the Disease
Brief Title: Brain Metastasis in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112951
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Cancer
Keywords: Breast Cancer; Treatment; Brain metastases; ErbB2 expression
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Brain Neoplasms | interventions — Trastuzumab; Lapatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women diagnosed with advanced breast cancer: Women diagnosed with advanced breast cancer during January 1, 1995-December 31, 2007 and treated as part of the Henry Ford Health System
  Interventions: Drug: Trastuzumab or Lapatinib

INTERVENTIONS:
Drug: Trastuzumab or Lapatinib — Anti-erbB2 therapy for breast cancer treatment will be analyzed as a class level variable; individual drugs including trastuzumab and lapatinib will also be explored as exposures if sufficient numbers of patients exist.

SUMMARY:
The purpose of this epidemiologic study is to establish a population-based cohort of women with advanced stage breast cancer which can be used to quantify the frequency and timing of brain metastases, and other distant metastases, in this patient population.

DETAILED DESCRIPTION:
A retrospective cohort study will be conducted in the Henry Ford Health System (HFHS). Using medical record review, we will identify all women diagnosed with advanced stage (stage III and IV) breast cancer between January 1, 1995- December 31, 2007. For each case included in the study, we will obtain data on demographics, tumor information, treatment related medical encounters and procedures, and occurrence and timing of brain and/or other distant metastases. The main outcome for this study is the development of distant metastases. Each patient in the cohort will be classified as to the occurrence and date of distant metastases. Metastases will be classified as Brain, Distant lymph node, Lung/pleural effusion, Liver, Bone, Other visceral, Other non-visceral.

Other secondary outcomes to be explored include:

* Survival after advanced breast cancer-time in months from the date of advanced stage breast cancer diagnosis until death or end of study period
* Time to brain metastases-time in month from the date of advanced stage breast cancer diagnosis until brain metastases diagnosis
* Survival after brain metastases-time in months from the date of diagnosis of brain metastases until death or end of study period

ELIGIBILITY:
Inclusion Criteria:

* Initially diagnosed with American Joint Commission on Cancer (AJCC) stage III or stage IV breast cancer between January 1, 1995 through December 31, 2007 -OR- diagnosed with AJCC stage I or II breast cancer and progressed to stage III or IV disease between January 1, 1995 through December 31, 2007;
* At least one year of follow-up after initial diagnosis (among patients who did not die before one year of follow-up); and
* Age 30 years or older at diagnosis.

Exclusion Criteria:

* Does not have at least one year of follow-up after initial diagnosis (among patients who did not die before one year of follow-up); and
* Age less than 30 years or older at diagnosis.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to retrospectively collect data on nearly 4,000 advanced breast cancer cases treated within the Henry Ford Health System
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Proportion of advanced stage breast cancer patients that develop brain metastases, overall and stratified by anti-HER2 therapy (for HER2+ patients only). | Time from breast cancer diagnosis until death or end of study periods (September 1, 2009)

SECONDARY OUTCOMES:
Overall survival from advanced stage breast cancer, overall and stratified by tumor characteristics and anti-HER2 therapy (for HER2+ patients only). | Time from diagnosis of advanced stage breast cancer until death or end of study period (September 1, 2009)
Time to brain metastases stratified by key tumor characteristics and anti-HER2 therapy (for HER2+ patients only). | Time from diagnosis of advanced stage breast cancer until brain metastases diagnosis
Survival after brain metastases diagnosis, overall and stratified by key tumor characteristics and anti-HER2 therapy (for HER2+ patients only) | Time from diagnosis of brain metastases until death or end of study period (September 1, 2009)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline